CLINICAL TRIAL: NCT06901544
Title: Capillary Leak Index as a Prognostic Indicator for Post-Operative Abdominal Sepsis in Critically Ill Patients
Acronym: CLI
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Osama Khalil, Principal Investigator, Ain Shams University
Other Study IDs: CLI In Abdominal sepsis
Record Dates: First submitted 2025-03-10; First posted 2025-03-30 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Intra-Abdominal Infections; Intestinal Obstruction; Appendicitis Acute; Perforated Viscus
Keywords: Capillary Leak Index; secondary abdominal sepsis; sepsis; Prognostic value; Good indicator; mortality; Intensive Care Unit; ICU
MeSH Terms: conditions — Intraabdominal Infections; Intestinal Obstruction; Appendicitis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low Capillary Leak Index < cutoff point 85.55: patient with Post operative Intra-abdominal sepsis with CLI at or less than 85.55 the cutoff point.
- high Capillary Leak Index > cutoff point 85.55: patient with Post operative Intra-abdominal sepsis with CLI higher than 85.55 the cutoff point.

SUMMARY:
In this study the investigators going to evaluate the "CLI" as an early prognostic indicator for post-operative abdominal sepsis in critically ill patients.

DETAILED DESCRIPTION:
Sepsis has been recognized as a life-threatening organ dysfunction caused by a dysregulated host response to infection. Considerable advances have since been made into the pathobiology (changes in organ function, morphology, cell biology, biochemistry, immunology, and circulation), management, and epidemiology of sepsis, suggesting the need for continuous research.

Peritonitis can be classified by the anatomical integrity of the abdominal cavity. Primary peritonitis is associated with undamaged intra-abdominal cavity organs. It is also known as spontaneous bacterial peritonitis and is treated without surgical intervention. The source of infection is often hard to establish and is usually found occurring in infants and cirrhotic patients.

Secondary peritonitis is an infection of the peritoneal cavity after hollow viscus perforation, anastomotic leak, ischemic necrosis, or other injuries of the gastrointestinal tract. Tertiary peritonitis is defined as a serious recurrent or persistent intra-abdominal infection after the successful control of secondary peritonitis. Irrespective of the cause, several measures are available and accepted as improving the survival rate, the most important being the early recognition of intra-abdominal infection. Efforts to achieve fluid balance should be initiated immediately to replace any intravascular insufficiency. Vasoactive agents may be necessary to augment and assist fluid restoration.

The treatment strategy for peritonitis primarily aims at the stabilization of possible organ dysfunction by routine intensive care medicine. Low risk secondary peritonitis (localized peritonitis), Ampicillin/Sulbactam or Carbapenem can be used as a monotherapy, however in combination therapy 2nd generation Cephalosporin + Metronidazole or 3rd generation Cephalosporin + Metronidazole can be used. High risk Secondary peritonitis Piperacillin/Tazobactam or Carbapenem or Tigecycline can be used as a monotherapy. A combination therapy 4th generation Cephalosporin + Metronidazole are usually used. Tertiary peritonitis antifungal therapy in high-risk patients and empirical therapy should cover the probable micro flora and should be changed according to the culture results.

Capillary leak syndrome (CLS) refers to a syndrome of deranged fluid homeostasis, often observed in critically ill patients, CLS is frequently defined by excessive fluid shift from the intravascular to the extravascular space, resulting in intravascular hypovolemia, extravascular edema formation, and hypo perfusion necessitating further fluid resuscitation. In health, fluid exchange between intravascular and extravascular spaces is vital for maintaining the body's homeostasis. However, disturbances in this delicate equilibrium, can lead to the clinical picture of CLS.

CLI is measured by dividing CRP level by albumin level. Systematic response to tissue injury, including major surgery, is marked by increased pro inflammatory cytokines, which promotes CRP production and capillary leakage. If the injury still exists, inflammatory process will continue.

Our study will be done to evaluate the association between capillary leak index (CLI) and intensive care unit (ICU) related mortality in patients underwent major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old presented with Post-operative intra-abdominal sepsis due to secondary peritonitis.
* Sex: Both sexes.
* Post-Operative secondary peritonitis eg. Perforated viscus and abdominal abscess.
* Estimated length of ICU stays ≥48 hrs.

Exclusion Criteria:

* Patient refusal.
* Advanced Liver diseases According New MELD score ≥ 20 )Kamath et al.,2001)
* Renal diseases (Moderate decrease in GFR 30-59 ml/min/1.73m²--Severe decrease in GFR 15-29 ml/min/1.73m²--Kidney failure less than 15 ml/min/1.73m² or on Hemodialysis).
* Pregnancy.
* Primary peritonitis.
* Tertiary peritonitis.
* Mortality within first 48hrs of ICU admission.
* Advanced malignancy ( Stage III localized malignancy with spreading lymph nodes Stage IV spreading to Other parts of the body such as to the liver, lungs and bones).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU Patient Post operative abdominal sepesis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Ahmed, MD., Study Director — Ain shams University Faculty of medicine; Hanaa A El-Gendy, MD, Study Chair — Ain Shams University Faculty of medicine
Locations (1):
- Surgical intensive Care Unit, Ain Shams University Hospitals., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Result] 12. Susanti A, Lestari MI, Sedono R, IA L. High capillary leak index is associated with increased risk of ICU-related mortality after major abdominal surgery. Critical Care & Shock. 2021 Nov 1;24(6).
- [Result] Sartelli M, Abu-Zidan FM, Catena F, Griffiths EA, Di Saverio S, Coimbra R, Ordonez CA, Leppaniemi A, Fraga GP, Coccolini F, Agresta F, Abbas A, Abdel Kader S, Agboola J, Amhed A, Ajibade A, Akkucuk S, Alharthi B, Anyfantakis D, Augustin G, Baiocchi G, Bala M, Baraket O, Bayrak S, Bellanova G, Beltran MA, Bini R, Boal M, Borodach AV, Bouliaris K, Branger F, Brunelli D, Catani M, Che Jusoh A, Chichom-Mefire A, Cocorullo G, Colak E, Costa D, Costa S, Cui Y, Curca GL, Curry T, Das K, Delibegovic S, Demetrashvili Z, Di Carlo I, Drozdova N, El Zalabany T, Enani MA, Faro M, Gachabayov M, Gimenez Maurel T, Gkiokas G, Gomes CA, Gonsaga RA, Guercioni G, Guner A, Gupta S, Gutierrez S, Hutan M, Ioannidis O, Isik A, Izawa Y, Jain SA, Jokubauskas M, Karamarkovic A, Kauhanen S, Kaushik R, Kenig J, Khokha V, Kim JI, Kong V, Koshy R, Krasniqi A, Kshirsagar A, Kuliesius Z, Lasithiotakis K, Leao P, Lee JG, Leon M, Lizarazu Perez A, Lohsiriwat V, Lopez-Tomassetti Fernandez E, Lostoridis E, Mn R, Major P, Marinis A, Marrelli D, Martinez-Perez A, Marwah S, McFarlane M, Melo RB, Mesina C, Michalopoulos N, Moldovanu R, Mouaqit O, Munyika A, Negoi I, Nikolopoulos I, Nita GE, Olaoye I, Omari A, Ossa PR, Ozkan Z, Padmakumar R, Pata F, Pereira Junior GA, Pereira J, Pintar T, Pouggouras K, Prabhu V, Rausei S, Rems M, Rios-Cruz D, Sakakushev B, Sanchez de Molina ML, Seretis C, Shelat V, Simoes RL, Sinibaldi G, Skrovina M, Smirnov D, Spyropoulos C, Tepp J, Tezcaner T, Tolonen M, Torba M, Ulrych J, Uzunoglu MY, van Dellen D, van Ramshorst GH, Vasquez G, Venara A, Vereczkei A, Vettoretto N, Vlad N, Yadav SK, Yilmaz TU, Yuan KC, Zachariah SK, Zida M, Zilinskas J, Ansaloni L. Global validation of the WSES Sepsis Severity Score for patients with complicated intra-abdominal infections: a prospective multicentre study (WISS Study). World J Emerg Surg. 2015 Dec 16;10:61. doi: 10.1186/s13017-015-0055-0. eCollection 2015. PMID 26677396
- [Result] Saravi B, Goebel U, Hassenzahl LO, Jung C, David S, Feldheiser A, Stopfkuchen-Evans M, Wollborn J. Capillary leak and endothelial permeability in critically ill patients: a current overview. Intensive Care Med Exp. 2023 Dec 20;11(1):96. doi: 10.1186/s40635-023-00582-8. PMID 38117435
- [Result] 9. PALACIOS MOGUEL, Paul et al. Capillary leak index as a new prognostic tool in septic shock Med. Crít. (Col. Mex. Med. Crít.) vol.32 no.3 Mexico City May/Jun. 2018.
- [Result] Meng R, Guan X, Sun L, Fei Z, Li Y, Luo M, Ma A, Li H. The efficacy and safety of eravacycline compared with current clinically common antibiotics in the treatment of adults with complicated intra-abdominal infections: A Bayesian network meta-analysis. Front Med (Lausanne). 2022 Sep 16;9:935343. doi: 10.3389/fmed.2022.935343. eCollection 2022. PMID 36186801
- [Result] Muresan MG, Balmos IA, Badea I, Santini A. Abdominal Sepsis: An Update. J Crit Care Med (Targu Mures). 2018 Oct 1;4(4):120-125. doi: 10.2478/jccm-2018-0023. eCollection 2018 Oct. PMID 30574564
- [Result] Morrissey I, Hackel M, Badal R, Bouchillon S, Hawser S, Biedenbach D. A Review of Ten Years of the Study for Monitoring Antimicrobial Resistance Trends (SMART) from 2002 to 2011. Pharmaceuticals (Basel). 2013 Nov 1;6(11):1335-46. doi: 10.3390/ph6111335. PMID 24287460
- [Result] Montravers P, Dufour G, Guglielminotti J, Desmard M, Muller C, Houissa H, Allou N, Marmuse JP, Augustin P. Dynamic changes of microbial flora and therapeutic consequences in persistent peritonitis. Crit Care. 2015 Mar 2;19(1):70. doi: 10.1186/s13054-015-0789-9. PMID 25887649
- [Result] Kamath PS, Wiesner RH, Malinchoc M, Kremers W, Therneau TM, Kosberg CL, D'Amico G, Dickson ER, Kim WR. A model to predict survival in patients with end-stage liver disease. Hepatology. 2001 Feb;33(2):464-70. doi: 10.1053/jhep.2001.22172. PMID 11172350
- [Result] Donnelly JP, Safford MM, Shapiro NI, Baddley JW, Wang HE. Application of the Third International Consensus Definitions for Sepsis (Sepsis-3) Classification: a retrospective population-based cohort study. Lancet Infect Dis. 2017 Jun;17(6):661-670. doi: 10.1016/S1473-3099(17)30117-2. Epub 2017 Mar 4. PMID 28268067
- [Result] Clements TW, Tolonen M, Ball CG, Kirkpatrick AW. Secondary Peritonitis and Intra-Abdominal Sepsis: An Increasingly Global Disease in Search of Better Systemic Therapies. Scand J Surg. 2021 Jun;110(2):139-149. doi: 10.1177/1457496920984078. Epub 2021 Jan 7. PMID 33406974
- [Result] 1. Ade Susanti1,2 , Mayang Indah Lestari et al. High capillary leak index is associated with increased risk of ICU-related mortality after major abdominal surgery Crit Care Shock 2021) 24:293-300.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: "100 Participants were recruited from Surgical intensive Care Unit, Ain Shams University Hospitals. In between March 2025 and Aug 2025." "Recruitment was conducted through ICU."
Pre-assignment Details: the 100 participants enrolled.
  * 50 participants of CLI at or less than of cutoff point 85.55 were enrolled.
  * 50 participants of CLI more than of cutoff point 85.55 were enrolled.
Groups:
- Low CLI at or Less Than Cutoff Point 85.55: 50 Participants patient with Post operative Intra-abdominal sepsis with CLI at or less than 85.55 the cutoff point.
  This group included 100 adult ICU patients with post-operative secondary intra-abdominal sepsis. The Capillary Leak Index (CLI) was calculated for each participant using the formula: (CRP ÷ Albumin) × 100. Patients were stratified into low and high CLI subgroups according to the cutoff Point of 85.55 for prognostic analysis.
- High CLI More Than Cutoff Point 85.55: 50 Participants patient with Post operative Intra-abdominal sepsis with High CLI more than 85.55 the cutoff point.
  This group included 100 adult ICU patients with post-operative secondary intra-abdominal sepsis. The Capillary Leak Index (CLI) was calculated for each participant using the formula: (CRP ÷ Albumin) × 100. Patients were stratified into low and high CLI subgroups according to the cutoff Point of 85.55 for prognostic analysis.
Period: Overall Study
Arm/Group | Low CLI at or Less Than Cutoff Point 85.55 | High CLI More Than Cutoff Point 85.55
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low CLI Equal or Less Than 85.55 Cutoff Point.: Adult ICU Patients with secondary peritonitis who had a baseline capillary leak index at or less than cutoff points 85.55 were enrolled with 48 hours of ICU admission and followed for 28 days mortality.
- High CLI Greater Than 85.55 Cutoff Point.: Adult ICU Patients with secondary peritonitis who had a baseline capillary leak index more than cutoff points 85.55 were enrolled with 48 hours of ICU admission and followed for 28 days mortality.
- Total: Total of all reporting groups
Arm/Group | Low CLI Equal or Less Than 85.55 Cutoff Point. | High CLI Greater Than 85.55 Cutoff Point. | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Mean (Full Range); unit: Age (years)]
  Age | 56 [18 to 88] | 60 [19 to 89] | 58 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 37 | 38 | 75
Diabetes mellitus disease (DM) [Count of Participants; unit: Participants] — patients with or without past medical history with Diabetes mellitus (DM)
  Participants
    positive | 14 | 18 | 32
    negative | 36 | 32 | 68
Cardiovascular diseases [Count of Participants; unit: Participants] — patients with or without Cardiovascular diseases
  Participants
    positive | 19 | 17 | 36
    negative | 31 | 33 | 64
Hepatic diseases [Count of Participants; unit: Participants] — according New MELD Score less than 20
  Participants
    Positive | 1 | 2 | 3
    Negative | 49 | 48 | 97
Renal diseases [Count of Participants; unit: Participants] — Mild GFR decrease (GFR > 60)
  Participants
    positive | 6 | 9 | 15
    negative | 44 | 41 | 85
surgical history [Count of Participants; unit: Participants] — history of surgical major operation
  Participants
    positive | 22 | 16 | 38
    negative | 28 | 34 | 62
Drugs History [Count of Participants; unit: Participants] — patient on regular medical Drugs intake for chronic diseases
  Participants
    positive | 27 | 24 | 51
    negative | 23 | 26 | 49
Acute Physiology and Chronic Health Evaluation (APACHE II),Sequential Organ Failure Assessment(SOFA) [Median (Inter-Quartile Range); unit: Score on a Scale] — * (APACHE II) score, a scale to scoring system for evaluating the severity of illness in patients admitted to an Intensive Care Unit (ICU) the score ranges from 0 to 71, with higher scores indicating greater disease severity and worse prognosis.
  * (SOFA score) a scale to scoring system used in intensive care units (ICUs) to objectively assess and monitor the severity of organ dysfunction and failure over time in critically ill patients Score ranges from 0 to 24 Higher SOFA scores indicate greater organ dysfunction and worse prognosis.
  Score on a Scale
    APACHE II Score | 19.5 [14.25 to 26.75] | 21.5 [16 to 29.75] | 20.5 [14.25 to 29.75]
    SOFA Score | 6.5 [4 to 9] | 10.5 [5 to 13.75] | 8.5 [4 to 13.75]
Abdominal Pain [Mean (Standard Deviation); unit: days]
  Pain Onset | 6.02 (4.44) | 5.5 (4.19) | 5.76 (4.3)
  Pain Duration | 6.28 (4.39) | 6.55 (4.75) | 6.42 (4.55)
GIT symptoms [Count of Participants; unit: Participants]
  positive | 32 | 18 | 50
  negative | 18 | 32 | 50
Kidney function tests [Mean (Full Range); unit: mg/dL] — laboratory investigation
  mg/dL
    Urea | 62.18 [19 to 379] | 85.1 [45 to 126] | 73.64 [19 to 379]
    Creatinine | 1.56 [0.4 to 14.5] | 2.53 [0.9 to 4.3] | 2.045 [0.4 to 14.5]
C Reactive Protein (CRP) [Mean (Full Range); unit: mg/dL] | 14.8 [1.6 to 32.4] | 31.11 [19.7 to 70] | 22.955 [1.6 to 70]
Fever [Count of Participants; unit: Participants]
  positive | 6 | 6 | 12
  negative | 44 | 44 | 88
Albumin [Mean (Full Range); unit: g/L] | 32.52 [21 to 48] | 26.62 [17 to 36] | 29.57 [17 to 48]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m2)] | 23.57 (2.84) | 24.16 (2.66) | 23.87 (2.75)
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died by Day 28
Description: Baseline CLI will be calculated on ICU admission . Mortality status (alive or dead) will be assessed at 28 days after ICU admission. The primary outcome is the number of participants who died from any cause by day 28 after ICU admission. The Association between basline CLI and 28-day all- cause mortality will be evaluated.
Time Frame: 28 days after ICU admission
Measure: Count of Participants; unit: Participants
Arm/Group | Low CLI equal or less than 85.55 cutoff point. | High CLI greater than 85.55 cutoff point.
Number analyzed (Participants) | 50 | 50
Participants | 8 [3 to 20] | 23 [2 to 16]
Statistical Analysis 1: Comparison: Low CLI equal or less than 85.55 cutoff point. vs High CLI greater than 85.55 cutoff point; Test type: Other — Comparison of 28-day mortality between groups using chi-squared test; p = 0.001, Chi-squared

2. Secondary Outcome: ICU Stay [Unit: More Than 3 Days].
Description: ICU Stay [Unit: more than 3 Days].
Time Frame: up to 28 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Low CLI equal or less than 85.55 cutoff point. | High CLI greater than 85.55 cutoff point.
Number analyzed (Participants) | 50 | 50
days | 7.96 [5 to 10] | 8.78 [7 to 12]
Statistical Analysis 1: Comparison: Low CLI equal or less than 85.55 cutoff point. vs High CLI greater than 85.55 cutoff point; Test type: Superiority; p = 0.243, t-test, 2 sided; Mean Difference (Final Values) = 0.243, 95% CI 2-sided [-0.567 to 2.207]

3. Secondary Outcome: Procalcitonin [Unit: ng/mL] [Time Frame: 3 Days]
Description: The Relationship Between Variables:
  The investigators will analyze CLI as a prognostic indicator using logistic regression to predict risk of ICU mortality.
Time Frame: up to 3 days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Low CLI equal or less than 85.55 cutoff point. | High CLI greater than 85.55 cutoff point.
Number analyzed (Participants) | 50 | 50
ng/ml | 8.65 (16.55) [0.05 to 90] | 16.62 (20.63) [0.05 to 86]
Statistical Analysis 1: Comparison: Low CLI equal or less than 85.55 cutoff point. vs High CLI greater than 85.55 cutoff point; Test type: Other — Comparison of mean PCT levels between groups using two-sample t-test; p = 0.037, t-test, 2 sided; Mean Difference (Final Values) = 7.97, 95% CI 2-sided [0.54 to 15.40]

ADVERSE EVENTS:
Time Frame: from the second day of ICU admission until end of follow-up, up to 28 days.
Description: "Adverse events were defined according to ClinicalTrials.gov standards. All participants were monitored daily during ICU stay and throughout the 28-day follow-up. Events were assessed by the study investigators and included in the analysis for the entire enrolled population."
Arm/Group | Low CLI Equal or Less Than 85.55 Cutoff Point. | High CLI Greater Than 85.55 Cutoff Point.
All-Cause Mortality (participants affected / at risk) | 8/50 | 23/50
Serious Adverse Events (participants affected / at risk) | 27/50 | 35/50
Other Adverse Events (participants affected / at risk) | 14/50 | 19/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low CLI Equal or Less Than 85.55 Cutoff Point. (N=50) | High CLI Greater Than 85.55 Cutoff Point. (N=50)
Disseminated intravascular coagulation (DIC) (Blood and lymphatic system disorders) | 1 (2) | 0 (0) — DIC occurs in severe form of sepsis complications.
Acute Kidney injury (AKI) (Renal and urinary disorders) | 15 (15) | 17 (17)
Multi Organ Disfunctions (General disorders) | 4 (4) | 6 (6)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low CLI Equal or Less Than 85.55 Cutoff Point. (N=50) | High CLI Greater Than 85.55 Cutoff Point. (N=50)
constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (16) | 7 (7)
fever (Immune system disorders) | 6 (6) | 10 (10)

LIMITATIONS AND CAVEATS:
In this study, 124 patients were assessed for eligibility, 18 patients did not meet the criteria and 6 patients refused to participate in the study. The remaining patients were randomly allocated into two equal groups (50 patients in each). All allocated patients were followed-up and analyzed statistically.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: plan of study (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT06901544/Prot_SAP_000.pdf